CLINICAL TRIAL: NCT06937294
Title: Metformin in Post Chronic Pancreatitis Diabetes Mellitus: a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Metformin in Post Chronic Pancreatitis Diabetes Mellitus
Acronym: MOOD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOOD202501
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to the experimental group (metformin) or the control group (placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a double-blind trail. Participants, investigators, care providers and outcomes assessors are blinded to the group allocations. Investigators and care providers provide guidance on drug use and lifestyle. Outcomes assessors are responsible for the follow-up of the patients. A study coordinator, who is not blinded to the group allocations, is appointed to oversee the coordination of the study and the maintenance of the blinding procedures. The study coordinator do not be allowed to communicate with others (participants, investigators, care providers and outcomes assessors) regarding the group allocations and clinical conditions of the participants. In the event of a serious adverse event, the blinding could be broken by contacting the study coordinator for safety considerations, and the reasons for unblinding were documented in detail.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Participants are administered metformin with an initial dose of 500 mg/day, which was incrementally increased by 500 mg/day each week until the maximum tolerated dose. The maximum dose of metformin is set at 2000 mg/day. After 2 weeks of administration, participants will undergo safety assessments, including complete blood count, urinalysis, liver function tests, and renal function tests. After attainment to a stable dose of metformin, participants will undergo follow-up assessments at 4 weeks, 8 weeks, and 12 weeks. The final evaluation of outcome measures will be completed at the 12-week follow-up.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Participants are administered a placebo, starting with one tablet per day, followed by an incremental increase of one tablet per week. In the absence of adverse reactions, the dosage is escalated up to a maximum of four tablets per day. After 2 weeks of administration, participants will undergo safety assessments, including complete blood count, urinalysis, liver function tests, and renal function tests. After attainment to a stable dose, participants will undergo follow-up assessments at 4 weeks, 8 weeks, and 12 weeks. The final evaluation of outcome measures will be completed at the 12-week follow-up.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Participants are administered metformin with an initial dose of 500 mg/day, which was incrementally increased by 500 mg/day each week until the maximum tolerated dose. The maximum dose of metformin is set at 2000 mg/day.
  Arms: Metformin
Drug: Placebo — Participants are administered a placebo, starting with one tablet per day, followed by an incremental increase of one tablet per week. In the absence of adverse reactions, the dosage is escalated up to a maximum of four tablets per day.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of metformin in treating patients with post chronic pancreatitis diabetes mellitus (PPDM-C). The main questions it aims to answer are:

* What is the efficacy of metformin in glycemic control in patients with PPDM-C?
* What is the incidence of adverse effects associated with metformin in patients with PPDM-C?

Participants will be randomly assigned to receive either metformin or a placebo to see if metformin provides significant glycemic control and to assess the safety profile of the treatment.

DETAILED DESCRIPTION:
Chronic pancreatitis (CP) is an irreversible chronic fibro-inflammatory disease caused by multiple factors. Patients often present with recurrent upper abdominal pain, dyspepsia, steatorrhea, and other symptoms. Typical imaging findings of CP include pancreatic duct calcification, ductal dilation, and parenchymal atrophy. As pancreatic fibrosis progresses, islet cells may also be damaged, leading to abnormal glucose metabolism or even diabetes mellitus (DM). Approximately 25-80% of CP patients develop DM which has been called post chronic pancreatitis diabetes mellitus (PPDM-C), with the prevalence increasing with the duration of CP. PPDM-C has garnered significant attention in the academic community due to its unique clinical manifestations and complications. However, there is currently no well-defined management strategy for PPDM-C.

The management of PPDM-C requires balancing pancreatic endocrine and exocrine functions, and developing individualized treatment strategies. Compared with T2DM patients, PPDM-C patients face greater difficulty in achieving optimal glycemic control. Currently, there is no standardized management for PPDM-C, with treatment protocol largely relying on clinical experience. Metformin is the most frequently used medication for PPDM patients (64.5%), and is typically the initial treatment. In PPDM-C patients, previous metformin use is associated with a survival benefit over those who have never used any antidiabetic drugs. However, there is lake of clinical trails specifically addressing PPDM-C to elucidate the the efficacy in glycemic control and safety of metformin.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years, any sex.
2. Patients diagnosed with chronic pancreatitis.
3. Diagnose diabetes at least 3 months after chronic pancreatitis diagnosis.
4. Never used any diabetes drug/glucose-lowering medication or had discontinued any glucose-lowering medications for at least 8 weeks prior to screening.
5. HbA1c criteria: 7.5%~9.0%.
6. BMI >18.5.
7. Provision of signed informed consent.

Exclusion Criteria:

1. Type 1 diabetes or secondary diabetes not caused by chronic pancreatitis (e.g. diabetes due to monogenic defects, cystic fibrosis, medications, autoimmune diseases, stress, or other factors).
2. Contraindications or history of intolerance or allergy to metformin.
3. Fasting C-peptide <0.3 nmol/L.
4. Acute episodes of chronic pancreatitis at enrollment or within 3 months prior to enrollment.
5. History of congestive heart failure (NYHA class 3 or greater), unstable angina, or other severe cardiovascular diseases.
6. History of cancer (except non-melanoma skin cancer) within 5 years prior to screening.
7. History of partial or total pancreatectomy.
8. History of or planning bariatric surgery.
9. Previous organ transplantation.
10. Treatment with oral or systemic glucocorticoids within 3 months prior to enrollment or plan to use during the study (inhaled steroids are permitted).
11. History of hemolytic anemia, chronic transfusion requirements, or other conditions rendering HbA1c results unreliable.
12. Other conditions requiring glucose-lowering medications, such as polycystic ovary syndrome.
13. Fasting blood glucose >11.1 mmol/L during screening, requiring immediate treatment as judged by the physician.
14. Sever psychiatric disorders or health conditions deemed unsuitable for clinical research participation.
15. Pregnancy or plans for pregnancy during the course of the study.
16. Any other condition considered by the investigator to be inappropriate for participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in glycosylated hemoglobin (HbA1c) | 12 weeks after the attainment of a stable dose
  The change in the value of glycosylated hemoglobin (HbA1c) collected at Week 12 (after the attainment of a stable does) relative to baseline.

SECONDARY OUTCOMES:
The proportion of patients with HbA1c below 6.5% at Week 12 | 12 weeks after the attainment of a stable dose
  At the Week 12 after the attainment of a stable does, the proportions of patients with glycosylated hemoglobin (HbA1c) levels exceeding 6.5% are assessed.
The proportion of patients with HbA1c below 7% at Week 12 | 12 weeks after the attainment of a stable dose
  At the Week 12 after the attainment of a stable does, the proportions of patients with glycosylated hemoglobin (HbA1c) levels exceeding 7% are assessed.
The proportion of patients with HbA1c below 7.5% at Week 12 | 12 weeks after the attainment of a stable dose
  At the Week 12 after the attainment of a stable does, the proportions of patients with glycosylated hemoglobin (HbA1c) levels exceeding 7.5% are assessed.
The incidence of adverse events | 12 weeks after the attainment of a stable dose
  Adverse events include hypoglycemia, diabetic ketoacidosis, hyperglycemic hyperosmolar state, acute pancreatitis and gastrointestinal symptoms (nausea, vomiting, diarrhea, etc.).
Blood glucose profile characteristics | 12 weeks after the attainment of a stable dose
  Blood glucose profile from continuous glucose monitoring system (CGMS) (unit: mmol/L or mg/dL).
Exploratory objectives: pancreatic and gut hormones | Baseline
  Levels of specific pancreatic hormones (C-peptide, insulin, glucagon, etc.) and gut hormones (ghrelin, gastric inhibitory peptide, glucagon like peptide-1, etc.) measured in venous blood (unit: mmol/L or mg/dL).
Exploratory objectives: pancreatic exocrine function | 12 weeks after the attainment of a stable dose
  Pancreatic exocrine function is evaluated by fecal elastase-1 test.
Exploratory objectives: scores of quality of life | 12 weeks after the attainment of a stable dose
  Quality of life scores for patients with chronic pancreatitis are obtained using SF-36 (36-Item Short Form Health Survey) which contains 8 dimensions scored from 0 to 100 (standardized converted scores). The higher score means better function.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, M.D., Study Chair — Changhai Hospital; Lianghao Hu, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cho J, Petrov MS. Pancreatitis, Pancreatic Cancer, and Their Metabolic Sequelae: Projected Burden to 2050. Clin Transl Gastroenterol. 2020 Nov;11(11):e00251. doi: 10.14309/ctg.0000000000000251. PMID 33259158
- [Result] Petrov MS. Diabetes of the exocrine pancreas: American Diabetes Association-compliant lexicon. Pancreatology. 2017 Jul-Aug;17(4):523-526. doi: 10.1016/j.pan.2017.06.007. Epub 2017 Jun 19. PMID 28655595
- [Result] Vege SS, Chari ST. Chronic Pancreatitis. N Engl J Med. 2022 Mar 3;386(9):869-878. doi: 10.1056/NEJMcp1809396. No abstract available. PMID 35235728
- [Result] Beyer G, Habtezion A, Werner J, Lerch MM, Mayerle J. Chronic pancreatitis. Lancet. 2020 Aug 15;396(10249):499-512. doi: 10.1016/S0140-6736(20)31318-0. PMID 32798493
- [Result] Pan J, Xin L, Wang D, Liao Z, Lin JH, Li BR, Du TT, Ye B, Zou WB, Chen H, Ji JT, Zheng ZH, Hu LH, Li ZS. Risk Factors for Diabetes Mellitus in Chronic Pancreatitis: A Cohort of 2,011 Patients. Medicine (Baltimore). 2016 Apr;95(14):e3251. doi: 10.1097/MD.0000000000003251. PMID 27057870
- [Result] Zhu X, Liu D, Wei Q, Lin H, Zhi M, Chen Y, Qi L, Waldron RT, Lugea A, Pandol SJ, Li L. New-Onset Diabetes Mellitus After Chronic Pancreatitis Diagnosis: A Systematic Review and Meta-analysis. Pancreas. 2019 Aug;48(7):868-875. doi: 10.1097/MPA.0000000000001359. PMID 31268977
- [Result] Olesen SS, Viggers R, Drewes AM, Vestergaard P, Jensen MH. Risk of Major Adverse Cardiovascular Events, Severe Hypoglycemia, and All-Cause Mortality in Postpancreatitis Diabetes Mellitus Versus Type 2 Diabetes: A Nationwide Population-Based Cohort Study. Diabetes Care. 2022 Jun 2;45(6):1326-1334. doi: 10.2337/dc21-2531. PMID 35312752
- [Result] Viggers R, Jensen MH, Laursen HVB, Drewes AM, Vestergaard P, Olesen SS. Glucose-Lowering Therapy in Patients With Postpancreatitis Diabetes Mellitus: A Nationwide Population-Based Cohort Study. Diabetes Care. 2021 Sep;44(9):2045-2052. doi: 10.2337/dc21-0333. Epub 2021 Aug 6. PMID 34362812
- [Result] Cho J, Scragg R, Pandol SJ, Goodarzi MO, Petrov MS. Antidiabetic Medications and Mortality Risk in Individuals With Pancreatic Cancer-Related Diabetes and Postpancreatitis Diabetes: A Nationwide Cohort Study. Diabetes Care. 2019 Sep;42(9):1675-1683. doi: 10.2337/dc19-0145. Epub 2019 Jun 21. PMID 31227582